CLINICAL TRIAL: NCT06971770
Title: EVALUATION OF SALIVARY HMGB1, sTREM-1 AND TNF-α LEVELS IN SMOKING AND NON-SMOKER INDIVIDUALS WITH DIFFERENT PERIODONTAL DISEASES
Brief Title: EVALUATION OF SALIVARY BİOMARKER LEVELS IN SMOKING AND NON-SMOKER INDIVIDUALS WITH DIFFERENT PERIODONTAL DISEASES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Berkay TAŞDEMİR, Research Assistant of Periodontology, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-TDU-DİŞF-0016
Record Dates: First submitted 2025-05-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases
Keywords: gingivitis; periodontitis; smoking; tnf-a; sTREM-1; HMGB-1
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Periodontitis; Smoking

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of saliva were obtained from systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20) and with 20 systemically healthy smoker individuals with periodontitis (PS, n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy periodontium (Experimental): Individuals who, in the evaluation made in 6 areas of each tooth, had bleeding on probing in less than 10% of the areas, had a probing depth of less than 4 mm and had no attachment loss.
  Interventions: Diagnostic Test: saliva obtaining
- gingivitis (Experimental): Individuals who have bleeding on probing in more than 10% of the areas, a probing depth of less than 4 mm and no attachment loss, based on an evaluation of 6 areas of each tooth.
  Interventions: Diagnostic Test: saliva obtaining
- non-smoker periodontitis (Experimental): Individuals who have bleeding on probing in 30% or more areas according to the evaluation made in 6 areas of each tooth, who have a probing pocket depth of 5 mm or more in at least 2 non-adjacent teeth in each quadrant of the jaw and who have attachment loss of 4 mm or more, and who have coronal 1/3 or more (horizontal and/or vertical) bone loss on radiographs.
  Interventions: Diagnostic Test: saliva obtaining
- smoker periodontitis (Experimental): Individuals who smoke at least 10 cigarettes a day, who have bleeding on probing in 30% or more areas according to the evaluation made in 6 areas of each tooth, who have a probing pocket depth of 5 mm or more in at least 2 non-adjacent teeth in each quadrant of the jaw and who have attachment loss of 4 mm or more, and who have coronal 1/3 or more (horizontal and/or vertical) bone loss on radiographs.
  Interventions: Diagnostic Test: saliva obtaining

INTERVENTIONS:
Diagnostic Test: saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
This study aimed to compare various cytokine levels in saliva samples in order to understand the pathogenesis of chronic inflammatory diseases. In particular, HMGB1, sTREM-1 and TNF-α levels were examined between smokers and non-smokers with periodontitis and non-smokers with gingivitis and periodontally healthy individuals. 80 systemically healthy individuals were included in the study. These individuals were divided into four groups: 20 non-smoker periodontally healthy, 20 non-smoker with gingivitis, 20 non- smokers with periodontitis and 20 smokers with periodontitis. Periodontal clinical parameters of each individual were measured and saliva samples were taken. HMGB1, sTREM-1 and TNF-α levels in the saliva samples were determined by enzyme-linked immunoassay (ELISA) method. Statistical analyses were performed on the data to examine the differences in cytokine levels between the groups and the relationships of these cytokines with clinical parameters. The findings obtained may contribute to the research of potential biomarkers that can be used in the diagnosis of periodontal diseases and new ways of treatment processes.

DETAILED DESCRIPTION:
This clinical study aims to comparatively investigate the salivary levels of HMGB1, sTREM-1, and TNF-α in individuals with periodontitis who smoke and do not smoke, as well as in non-smoking individuals with gingivitis and periodontal health. Based on the results, the study seeks to determine the diagnostic potential of these cytokines in periodontal disease and the effect of smoking on their levels.

Periodontal disease is a multifactorial condition characterized by inflammation of the periodontal tissues, associated with plaque biofilms and mediated by the host response, leading to progressive loss of supporting structures and periodontal attachment. Gingivitis is defined as plaque-induced inflammation of the gingival tissues without loss of attachment. It is a reversible condition that typically resolves within approximately one week following the implementation of oral hygiene measures. It is widely accepted that untreated gingival lesions may progress to periodontitis in susceptible individuals. The transition from gingivitis to periodontitis occurs with the destruction of periodontal ligament fibers and alveolar bone. The most significant predisposing factor for periodontitis is poor oral hygiene, as the primary trigger of periodontitis lesions is microbial dental plaque, which contains numerous pathogenic bacteria. Among these, the red complex-Porphyromonas gingivalis, Tannerella forsythia, and Treponema denticola-poses the highest risk for the development of active periodontitis lesions.

Although the pathogenesis of periodontitis is not fully understood, it is well established that tissue destruction is largely due to the host immune response against bacteria and their by-products in dental plaque. The host-pathogen interaction triggers a cascade of immunoinflammatory events, leading to excessive release of proinflammatory cytokines such as interleukin-1 (IL-1), IL-6, prostaglandin E2 (PGE2), and tumor necrosis factor-α (TNF-α), as well as endopeptidases such as matrix metalloproteinases (MMPs), resulting in periodontal breakdown. Inflammation in both localized inflammatory lesions like periodontitis and systemic connective tissue diseases involving multiple tissues and organs is associated with increased levels of cytokines, prostaglandins, and MMPs in affected tissues and systemic circulation.

The available data indicate that periodontal disease exhibits a dynamic pattern of exacerbation and remission characterized by progression and regression of the disease. Different regions in the oral cavity display variable rates of attachment loss, and these regions appear to arise randomly. Active periodontal disease sites are believed to be associated with alterations in the inflammatory cell population, characterized by a significantly higher presence of mast cells, monocytes/macrophages, and plasma cells compared to inactive sites. These cells contribute to the activation and expression of proinflammatory mediators such as IL-1, IL-6, and TNF-α via stimulation of monocytes/macrophages, lymphocytes, fibroblasts, and other related cellular elements. These cytokines and inflammatory mediators promote alveolar bone resorption and collagen degradation, primarily through matrix metalloproteinases, which play a crucial role in tissue destruction associated with periodontal activity.

High mobility group box (HMGB) proteins are non-histone nuclear proteins with various intracellular functions. Initially isolated from the nucleus in the 1970s, they were named for their rapid migration in sodium dodecyl sulfate polyacrylamide gel electrophoresis. The HMGB family includes HMGB1, HMGB2, and HMGB3. While HMGB2 and HMGB3 exhibit limited expression, HMGB1 is widely expressed and its expression is regulated by environmental factors. HMGB1 plays a role in both acute and chronic inflammatory responses, as well as in wound healing. Secreted by activated macrophages, HMGB1 can activate other immune cells, acting as a cytokine. HMGB1 also promotes macrophage activation through HMGB1/RAGE interaction, JNK (c-Jun N-terminal kinase) activation, and upregulation of caspase-3 and caspase-9. Extracellular HMGB1 transmits inflammatory signals by binding to receptors such as RAGE (receptor for advanced glycation end products), TLR-2, TLR-4, and TLR-9. These receptors are believed to play a role in inflammatory processes. HMGB1 is involved in various acute and chronic inflammatory conditions, including rheumatoid arthritis, osteoarthritis, cancer, lupus, and periodontitis. However, only a limited number of studies have investigated the role of HMGB1 in the pathogenesis of periodontitis. Compared to inflamed gingival tissue, higher concentrations of HMGB1 have been detected in gingival crevicular fluid (GCF). Additionally, HMGB1 mRNA and protein levels are highly induced in mouse periodontal ligament fibroblasts stimulated with lipopolysaccharide (LPS) and interleukin-1β. In experimental models, elevated HMGB1 levels, in combination with IL-1β and TNF-α, contribute to alveolar bone loss in periodontitis, suggesting a role for HMGB1 in the disease. However, the mechanism by which HMGB1 contributes to periodontitis and peri-implant diseases, as well as the effect of smoking on salivary HMGB1 levels, remains unclear.

Triggering receptor expressed on myeloid cells-1 (TREM-1) is a recently identified molecule expressed on neutrophils and macrophages, known to amplify the inflammatory response. In humans, the TREM gene family includes TREM-1 and TREM-2 on chromosome 6q21, whereas TREM-3, a pseudogene in humans, is functional in mice. TREM-1 is a transmembrane protein with extracellular, transmembrane, and short cytoplasmic domains. A notable feature of the TREM family is the ability to be released in a soluble form. Soluble TREM-1 (sTREM-1) has been identified in the plasma and biological fluids of patients and animals with various infections and diseases. It is detectable in culture supernatants of mononuclear phagocytes stimulated with LPS, in the plasma of humans administered LPS, in the plasma of endotoxemic mice, in the plasma of septic patients, and in the bronchoalveolar lavage (BAL) fluid of pneumonia patients. TREM-1 is a novel receptor of the immunoglobulin superfamily expressed on the surface of monocytes, macrophages, and neutrophils and is a key regulator of innate immunity. It plays a critical role in amplifying the inflammatory cytokine response induced by LPS and other microbial products. sTREM-1 is released from cells and has been reported as a useful diagnostic marker in body fluids. Recent studies have shown elevated serum sTREM-1 levels in patients with inflammatory bowel disease and ankylosing spondylitis. In vitro studies have demonstrated that P. gingivalis induces TREM-1 expression in monocytes, facilitates its conversion to sTREM-1, and is accompanied by increased production of proinflammatory cytokines. Interestingly, these effects can be abolished by doxycycline. Recent clinical studies have reported higher sTREM-1 levels in gingival crevicular fluid from periodontitis sites compared to healthy sites and in the saliva of periodontitis patients compared to non-periodontitis individuals. However, the differences in salivary sTREM-1 levels between periodontitis and gingivitis forms, as well as between smoking and non-smoking periodontitis cases, remain unclear.

Tumor necrosis factor-alpha (TNF-α) is a 26 kDa membrane-bound cytokine that mediates the inflammatory response. It is a major mediator of the acute inflammatory response to Gram-negative bacteria and other microorganisms and is responsible for many systemic complications during infection. TNF-α plays critical roles in anti-tumor activity, immune modulation, inflammation, anorexia, septic shock, viral replication, and hematopoiesis. The principal cellular source of TNF-α is activated mononuclear phagocytes, although activated T cells, NK cells, and mast cells also produce TNF. LPS is the strongest inducer of TNF secretion by macrophages. Interferon-gamma (IFN-γ), produced by T cells and NK cells, enhances LPS-induced TNF production. TNF-α functions by promoting the recruitment of neutrophils and monocytes to sites of infection by inducing the release of adhesion molecules from vascular endothelial cells and leukocytes, facilitating leukocyte adhesion to the endothelium. It also induces chemokine release from endothelial cells and macrophages, promoting chemotaxis and accumulation of leukocytes at the site of infection. In severe infections, excessive TNF production can result in systemic clinical and pathological abnormalities. If the stimulus is particularly strong, TNF may enter the bloodstream and act as an endocrine hormone. TNF also enhances IL-1 production in mononuclear phagocytes and stimulates the differentiation of osteoclast precursors, contributing to bone resorption. Additionally, TNF-α induces apoptosis in fibroblasts, thereby limiting tissue repair. As a potent inflammatory mediator, TNF-α plays a significant role in the pathogenesis of periodontitis, a disease characterized by inflammation. It has also been reported to contribute to bone resorption. TNF-α stimulates gingival fibroblasts to produce collagenase, leading to tissue destruction. In studies evaluating the role of IL-1 and TNF-α in periodontal inflammation and bone loss, the administration of their inhibitory receptors in animal models resulted in a 60-80% reduction in inflammatory cells near bone, osteoclast formation, and bone loss.

According to 2015 WHO data, approximately 1.1 billion people worldwide use tobacco products. Due to its high nicotine content, tobacco has a strong potential for addiction. Tobacco products contain more than 4,000 chemicals, with tar, a carcinogen, and nicotine, the addictive component, being the most harmful. The impact of smoking varies based on the age of smoking initiation, duration, daily consumption, form of use, and tar/nicotine content of the cigarette. While the primary effect of smoking is on the respiratory system, it also negatively affects the circulatory, digestive, nervous, and immune systems. Literature indicates that smoking is an important environmental risk factor in the pathogenesis and progression of periodontal disease. Smoking contributes to periodontal tissue destruction via multiple mechanisms, including alterations in microcirculation, host immune response, connective tissue, and bone metabolism. It is recognized as an independent risk factor for the onset and progression of periodontal disease. Cross-sectional and longitudinal studies provide strong evidence that smoking increases the risk of developing periodontal disease. Compared to non-smokers, smokers exhibit higher prevalence and severity of periodontitis, earlier onset, faster progression, and poorer response to periodontal treatment. Despite higher plaque scores in smokers, reduced gingival bleeding has been reported. Smoking negatively affects both the local and systemic health of periodontal tissues and host responses. It reduces phagocytosis and chemotaxis of peripheral blood neutrophils and allows nicotine migration to oral PMNLs. Nicotine, the most common compound found in tobacco products, inhibits the production of superoxide and IL-1β, thereby impairing the defensive functions of neutrophils and monocytes. This impairment of aerobic antimicrobial function may promote microbial changes in the subgingival environment.

Saliva is an extracellular fluid containing various components such as electrolytes, epithelial cells, antibacterial compounds, and enzymes. Several studies have highlighted the potential diagnostic value of salivary analyses. Investigations into the risk factors and biomarkers of periodontal infections may benefit from the simple and rapid method of saliva sampling. According to current knowledge, no studies have yet evaluated and compared HMGB1, sTREM-1, and TNF-α levels in saliva samples in the context of both periodontal disease and smoking. This study aims to analyze the salivary levels of HMGB1, sTREM-1, and TNF-α in systemically healthy individuals with periodontal health, gingivitis, and periodontitis (with and without smoking), to investigate their changes in relation to disease presence and smoking, their association with clinical parameters, and to determine their diagnostic potential or possible therapeutic implications through their signaling pathways.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (Determination of volunteers will be based on patient statements in the anamnesis. No additional examination will be performed.)
* At least 16 permanent teeth in the mouth
* For non-smoking groups: never smoked
* For the smoking group: smoking at least 10 cigarettes per day
* No continuously used medications
* No use of antibiotics, anti-inflammatory drugs, and systemic corticosteroids in the last 6 months
* Not pregnant or breastfeeding
* No periodontal treatment in the last 6 months
* For the Periodontitis group: based on the evaluation of 6 sites per tooth, ≥30% bleeding on probing, probing depth ≥5 mm and clinical attachment loss ≥4 mm in at least 2 non-adjacent teeth in a quadrant, and radiographic bone loss of coronal 1/3 or more (horizontal and/or vertical)
* For the Gingivitis group: based on the evaluation of 6 sites per tooth, ≥10% bleeding on probing, probing depth <4 mm, and no clinical attachment loss
* For the Healthy group: based on the evaluation of 6 sites per tooth, <10% bleeding on probing, probing depth <4 mm, and no clinical attachment loss.

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Salivary TNF-α levels | 24 hours after taking the clinical measurements at the first visit
  the total amount of TNF-α in saliva
Salivary sTREM-1 level | 24 hours after taking the clinical measurements at the first visit
  the total amount of sTREM-1 in saliva
Salivary HMGB-1 levels | 24 hours after taking the clinical measurements at the first visit
  the total amount of HMGB-1 in saliva

SECONDARY OUTCOMES:
Probing Depth | during the initial visit
  With the help of a periodontal probe, the distance between the gingival margin and the sulcus/pocket base will be measured from six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. During the measurement, care will be taken to ensure that the probe is parallel to the long axis of the tooth and that excessive force is not applied. The values will be summed and divided by 6 to calculate the average PD for each patient.
clinical attachment level | during the initial visit
  With the help of a periodontal probe, the distance between the enamel-cement border and the sulcus/pocket base will be measured at six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. The values will be summed and divided by 6 to calculate the average amount of clinical attachment level for each patient.
Plaque Index | during the initial visit
  For Silness&Löe plaque index measurement, values will be obtained from four surfaces of each tooth: mesial, distal, vestibular and palatinal. The values will be summed and divided by four to determine the PI score for each tooth. Scoring will be done as follows; 0: No bacterial plaque on the gingival area of the tooth surface. 1: No bacterial plaque is visible on the surface of the tooth by eye, but after probing, bacterial plaque is observed at the tip of the probe. 2: The gingival area is covered with a thin to moderate amount of bacterial plaque, which is visible by eye. 3: There is a large amount of soft debris, the thickness of which completely fills the gingival groove and the interdental space is filled with soft debris
gingival index | during the initial visit
  According to Löe&Silness gingival index; vestibule, lingual, mesial and distal surfaces of all teeth will be examined. The values will be summed and divided by four to determine the GI score for each tooth. 0: Healthy gingiva. 1: Mild inflammation, mild discoloration and edema but no bleeding after probing. 2: Moderate inflammation, edema, redness and brightness, bleeding on probing. 3: Severe inflammation and redness, edema, ulceration and tendency to spontaneous bleeding.
bleeding on probing | during the initial visit
  The following index criteria will be used to determine the degree of inflammation in the soft tissue surrounding the vestibular, lingual, mesial and distal surfaces of all teeth. The number of positive (+) scoring areas on the examined surfaces will be calculated as a percentage of the total number of examined areas. (-): No bleeding when the periodontal probe is passed along the gingival sulcus. (+): Bleeding is present at the gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No